CLINICAL TRIAL: NCT01091636
Title: Randomized Trial of Intraoperative Hyperthermic Intraperitoneal Chemotherapy Followed by Intravenous Chemotherapy in Patients With Ovarian Cancer
Brief Title: Intraoperative Hyperthermic Intraperitoneal Chemotherapy With Ovarian Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Ajou University (Other)
Responsible Party: Principal Investigator, Sang-Yoon Park, Gynecologic Oncologist, Center for Gynecologic Cancer, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCCCTS-06-222
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Intervention Model Description: HIPEC vs. no HIPEC after primary cytoreductive surgery or interval cytoreductive surgery
Who Masked: Participant
Masking Description: Blinded to the participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIPEC (Experimental): Intraoperative Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in Patients with Ovarian Cancer after primary cytoreductive surgery or interval cytoreductive surgery
  Interventions: Procedure: Hyperthermic Intraperitoneal Chemotherapy
- No HIPEC (No Intervention): Primary cytoreductive surgery or interval cytoreductive surgery

INTERVENTIONS:
Procedure: Hyperthermic Intraperitoneal Chemotherapy — 41.5 oC injected into the perfusion cisplatin (75 mg/m2)during 90min
  Other Names: Belmont Instrument Corporation
  Arms: HIPEC

SUMMARY:
The current standard treatment for ovarian cancer, tubal cancer, and primary peritoneal cancer is maximal cytoreductive surgery followed by chemotherapy. Recent randomized trials of Gynecologic Oncology Group (GOG) revealed the survival gain in intraperitoneal chemotherapy compared to the intravenous chemotherapy after the optimal cytoreduction in ovarian cancer (GOG#104, GOG#114, GOG#172). Experts attributed such survival gain to the earlier cycles of intraperitoneal chemotherapy when adhesion was minimal from extensive cytoreductive procedures.

Hyperthermia has an anti-cancer activity itself. Especially, hyperthermia promotes chemotherapy to penetrate deeper into the cancer tissue. Therefore, the combination of intraperitoneal chemotherapy with hyperthermia theoretically could lead to higher response rate and better survival outcomes.

*HIPEC: hyperthermic intraperitoneal chemotherapy

There will be an interim analysis when 50% of patients are enrolled.

At the interim analysis, a statistical test will be performed. The nominal significance levels will be determined later. The exact nominal significance level will be determined based on the exact number of events at the time of the interim analysis. The Stopping boundaries will be calculated using an O'Brien-Fleming error spending function

DETAILED DESCRIPTION:
If a patient is allocated to operation to remove ovarian cancer and metastatic disease in the abdomen, this trial could be considered. Before operation, laboratory test results, image result, patient's medical history, and baseline quality of life will be checked and reviewed.

When optimal cytoreduction (residual tumor<1cm) is attained, this HIPEC (hyperthermic intraperitoneal chemotherapy) could be considered. For the primary advanced epithelial ovarian cancer, HIPEC will be performed at random. For the recurrent ovarian cancer, HIPEC will be performed after completion of cytoreductive procedures. Usually, HIPEC takes one and half hours after cytoreductive surgery.

After cytoreductive surgery followed by HIPEC, adjuvant chemotherapy will be added. The cycle of chemotherapy will be determined according to the patients' clinical outcomes. The laboratory test results, image result, patient's medical history, and baseline quality of life will be checked after the operation, during chemotherapy, and after chemotherapy.

Cytoreduction: an operation to remove ovarian cancer and its metastatic disease

There will be an interim analysis when 50% of patients are enrolled.

At the interim analysis, a statistical test will be performed. The nominal significance levels will be determined later. The exact nominal significance level will be determined based on the exact number of events at the time of the interim analysis. The Stopping boundaries will be calculated using an O'Brien-Fleming error spending function

ELIGIBILITY:
Inclusion Criteria:

1. Disease status Primary ovarian cancer, tubal cancer, and primary peritoneal cancer (Stage III or more)
2. Residual tumor < 1cm after completion of cytoreductive surgery
3. Age < 75 year
4. Expected survival > 3 months
5. Performance status: ECOG 0-1
6. Adequate bone marrow function Hb ≥8 g/dl (After correction in case of iron deficient anemia) WBC ≥ 3,000/mm3, Platelet ≥ 100,000/mm3
7. Adequate renal function Creatinine ≤ 1.5 mg/dl
8. Adequate hepatic function Bilirubin ≤ 1.5 mg/dl and AST and ALT ≤ 80 IU/L
9. Optimal cardiopulmonary function for surgery
10. Voluntary participation after getting written informed consent.

Exclusion Criteria:

1. Unresectable extraperitoneal metastasis (brain, bone, lung parenchyme, and supraclavicular lymph node)
2. Suboptimal debulking (residual tumor > 1cm)
3. Previous History of other malignancies (except excision of skin cancer, thyroid cancer)
4. Serious heart disease or renal failure
5. Serious cardiopulmonary insufficiency
6. Uncontrolled infection
7. Uncontrolled intercurrent disease
8. Psychogenic disorder
9. Patients who are suitable candidates by legally
10. Pregnant or breast-feeding patients
11. Patients who are unsuitable candidates by doctor's decision
12. MMMT
13. Cancer tissue is not confirmed during surgery after neo-adjuvant chemotherapy

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2010-03; Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 2 years
  To assess progression free survival rate during 2 years after Intraoperative Hyperthermic Intraperitoneal Chemotherapy followed by Intravenous Chemotherapy in Patients with Ovarian Cancer.

SECONDARY OUTCOMES:
Overall survival, quality of life | 3 years
  Ovarian cancer patients after HIPEC are observed complication and 3-year survival rate.
  Ovarian cancer patients after HIPEC are analyzed quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Yoon Park, MD, Ph.D., Principal Investigator — National Cancer Center in Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lim MC, Kang S, Choi J, Song YJ, Park S, Seo SS, Park SY. Hyperthermic intraperitoneal chemotherapy after extensive cytoreductive surgery in patients with primary advanced epithelial ovarian cancer: interim analysis of a phase II study. Ann Surg Oncol. 2009 Apr;16(4):993-1000. doi: 10.1245/s10434-008-0299-y. Epub 2009 Jan 24. PMID 19169758
- [Derived] Kim JH, Chun SY, Lee DE, Woo YH, Chang SJ, Park SY, Chang YJ, Lim MC. Cost-effectiveness of hyperthermic intraperitoneal chemotherapy following interval cytoreductive surgery for stage III-IV ovarian cancer from a randomized controlled phase III trial in Korea (KOV-HIPEC-01). Gynecol Oncol. 2023 Mar;170:19-24. doi: 10.1016/j.ygyno.2022.12.021. Epub 2023 Jan 4. PMID 36608383
- [Derived] Kim JH, Lee DE, Lee Y, Ha HI, Chang YJ, Chang SJ, Park SY, Lim MC. Quality of life outcomes from the randomized trial of hyperthermic intraperitoneal chemotherapy following cytoreductive surgery for primary ovarian cancer (KOV-HIPEC-01). J Gynecol Oncol. 2022 Jul;33(4):e54. doi: 10.3802/jgo.2022.33.e54. Epub 2022 May 31. PMID 35712968
- [Derived] Lim MC, Chang SJ, Park B, Yoo HJ, Yoo CW, Nam BH, Park SY; HIPEC for Ovarian Cancer Collaborators. Survival After Hyperthermic Intraperitoneal Chemotherapy and Primary or Interval Cytoreductive Surgery in Ovarian Cancer: A Randomized Clinical Trial. JAMA Surg. 2022 May 1;157(5):374-383. doi: 10.1001/jamasurg.2022.0143. PMID 35262624